CLINICAL TRIAL: NCT06848699
Title: A Phase Ib/ II Clinical Study to Evaluate the Safety ,Torlerbility , and Efficacy of HLX43 (Anti-PD-L1 ADC) in Combination With Serplulimab (Anti-PD-1 Humanized Monocl ) in Patients With Advanced/Metastatic Solid Tumors
Brief Title: A Phase Ib/II Clinical Study to Evaluate HLX43 in Combination With Serplulimab in Patients With Advanced/Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HLX43HLX10-ST201
Record Dates: First submitted 2025-01-22; First posted 2025-02-27 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Solid Tumor Cancer; Non Small Cell Lung Cancer
Keywords: HLX43
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- HLX43 dose 1 (Experimental): Patients with good tolerability and well controlled disease will receive the treatment once every 3 weeks (Q3W), Until disease progression, initiation of a new anti-tumor therapy, death, emergence of intolerable toxicity, or withdrawal of informed consent (whichever occurs first)
  Interventions: Drug: HLX43 dose 1; Drug: Serplulimab
- HLX43 dose 2 (Experimental): : Patients with good tolerability and well controlled disease will receive the treatment once every 3 weeks (Q3W), Until disease progression, initiation of a new anti-tumor therapy, death, emergence of intolerable toxicity, or withdrawal of informed consent (whichever occurs first)
  Interventions: Drug: HLX43 dose 2; Drug: Serplulimab
- HLX43 dose 3 (Experimental): : Patients with good tolerability and well controlled disease will receive the treatment once every 3 weeks (Q3W), Until disease progression, initiation of a new anti-tumor therapy, death, emergence of intolerable toxicity, or withdrawal of informed consent (whichever occurs first)
  Interventions: Drug: HLX43 dose 3; Drug: Serplulimab
- HLX43 dose 4 (Experimental): : Patients with good tolerability and well controlled disease will receive the treatment once every 3 weeks (Q3W), Until disease progression, initiation of a new anti-tumor therapy, death, emergence of intolerable toxicity, or withdrawal of informed consent (whichever occurs first)
  Interventions: Drug: HLX43 dose 4; Drug: Serplulimab
- HLX43 dose 5 (Experimental): Patients with good tolerability and well controlled disease will receive the treatment once every 3 weeks (Q3W), Until disease progression, initiation of a new anti-tumor therapy, death, emergence of intolerable toxicity, or withdrawal of informed consent (whichever occurs first)
  Interventions: Drug: HLX43 dose 5; Drug: Serplulimab

INTERVENTIONS:
Drug: HLX43 dose 1 — HLX43 is an anti-PD-L1 monoclonal antibody conjugated with a novel high potency DNA topoisomerase I (topo I) inhibitor, with a drug-antibody-ratio (DAR) of 8.
  Arms: HLX43 dose 1
Drug: HLX43 dose 2 — HLX43 is an anti-PD-L1 monoclonal antibody conjugated with a novel high potency DNA topoisomerase I (topo I) inhibitor, with a drug-antibody-ratio (DAR) of 8.
  Arms: HLX43 dose 2
Drug: HLX43 dose 3 — HLX43 is an anti-PD-L1 monoclonal antibody conjugated with a novel high potency DNA topoisomerase I (topo I) inhibitor, with a drug-antibody-ratio (DAR) of 8.
  Arms: HLX43 dose 3
Drug: HLX43 dose 4 — HLX43 is an anti-PD-L1 monoclonal antibody conjugated with a novel high potency DNA topoisomerase I (topo I) inhibitor, with a drug-antibody-ratio (DAR) of 8.
  Arms: HLX43 dose 4
Drug: HLX43 dose 5 — HLX43 is an anti-PD-L1 monoclonal antibody conjugated with a novel high potency DNA topoisomerase I (topo I) inhibitor, with a drug-antibody-ratio (DAR) of 8.
  Arms: HLX43 dose 5
Drug: Serplulimab — anti-PD-1 humanized monoclonal antibody injection

SUMMARY:
The study is being conducted to explore the reasonable dosage and evaluate the efficacy, safety and tolerability of HLX43 (Anti-PD-L1 ADC) in combination with Serplulimab (anti-PD-1 humanized monoclonal antibody injection) in patients with advanced/metastatic solid tumors

DETAILED DESCRIPTION:
This study is an open-label phase Ib/II clinical study to explore the reasonable dosage and evaluate the efficacy, safety and tolerability of HLX43 (Anti-PD-L1 ADC) in combination with Serplulimab (anti-PD-1 humanized monoclonal antibody injection) in Patients with advanced/metastatic solid tumors. The study is divided into two phases: phase Ib dose escalation and phase II dose expansion.The subjects will receive different dosages of HLX43 combined with a fixed dosage (300 mg) of serplulimab, administered via intravenous infusion every 3 weeks (Q3W) .

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participate in the clinical trial; fully understand and be informed about this study and sign the Informed Consent Form (ICF); be willing and able to comply with and complete all trial procedures;
2. Age at the time of signing the ICF is ≥ 18 years and ≤ 75 years;
3. Phase Ib enrollment of patients with histologically or cytologically confirmed advanced /metastatic solid tumor who have experienced treatment failure or for whom no standard treatment is available;Phase II enrollment includes advanced /metastatic NSCLC subjects confirmed by histology or cytology, requiring the presence of EGFR mutation and failure or intolerance to EGFR-TKI or/and platinum-based chemotherapy.
4. Within 4 weeks prior to the first dose, at least one measurable lesion assessed by the investigator according to RECIST 1.1;
5. Subjects must provide qualified tumor tissue samples for the determination of PD-L1 expression levels.
6. The ECOG PS score within 7 days prior to the first use of the Investigational Product is 0 or 1;
7. Expected survival ≥ 12 weeks;
8. Major organ functions are normal, meeting the following criteria (within 14 days prior to the first administration in this study, no transfusion, albumin, recombinant human thrombopoietin, or colony-stimulating factor (CSF) treatment was received):
9. Female subjects of childbearing potential must meet the following criteria:

   a)The blood pregnancy test must be negative within 7 days prior to the first administration of the medication; b)Agree to use at least one highly effective method of contraception during the trial period and for at least 6 months after the last administration of the drug;c)Breastfeeding is contraindicated.
10. Male subjects must meet the following criteria: agree to use at least one highly effective method of contraception during the trial and for at least 6 months after the last dose.

Exclusion Criteria:

1. History of any second malignancy within 3 years prior to randomization, except for early-stage malignancies (carcinoma in situ or stage I tumors) that have received radical treatment, such as non-melanoma skin cancer, cervical carcinoma in situ, localized prostate cancer, ductal carcinoma in situ of the breast, and papillary thyroid carcinoma.
2. Previously experienced ≥ Grade 3 immune-related Adverse Events during immunotherapy.
3. Pleural effusion or pericardial effusion, or ascites requiring clinical intervention as determined by the investigator;
4. Subjects with clinical symptoms of brain metastases, spinal cord compression, meningitis carcinomatosa, or other evidence indicating that brain or spinal cord metastatic lesions are not yet controlled; Note: Subjects with asymptomatic or stable brain metastases, spinal cord compression, or meningitis carcinomatosa as determined by theinvestigator may be eligible for enrollment;
5. Subjects with a history or current condition of interstitial pneumonia, pneumoconiosis, radiation pneumonitis, drug-related pneumonia, or severe impairment of pulmonary function, as determined by the sub investigator, that may interfere with the detection and management of suspected drug-related pulmonary toxicity;
6. The subject has poorly controlled cardiovascular and cerebrovascular clinical symptoms or diseases, including but not limited to: (1) NYHA class II or higher heart failure or left ventricular ejection fraction (LVEF) <50%; (2) unstable angina; (3) myocardial infarction or cerebrovascular accident within the past 6 months (excluding lacunar infarction, minor cerebral ischaemia, or transient ischaemic attack); (4) uncontrolled arrhythmia (including QTc interval ≥450 ms for males and ≥470 ms for females, with QTc interval calculated using the Fridericia formula); (5) poorly controlled hypertension (systolic blood pressure >150 mmHg and/or diastolic blood pressure >100 mmHg despite active treatment);
7. History of immunodeficiency diseases, including testing positive for human immunodeficiency virus (HIV), or having other acquired or congenital immunodeficiency diseases, or a history of organ transplant;
8. Has active pulmonary tuberculosis;
9. Subjests with active HBV, HCV infection or co-infection;
10. There is a known active or suspected autoimmune disease. Enrollment is allowed for subjects in a stable condition who do not require systemic immunosuppressive therapy.
11. Subjects requiring systemic corticosteroids (>10 mg/day prednisone therapeutic dosage) or other immunosuppressive drug therapy within 14 days prior to the first administration of the Investigational Product or during the study. However, the following situations allow for enrollment: in the absence of active autoimmune disorders, the use of topical external application or inhaled steroids and adrenal hormone replacement therapy at a dosage ≤10 mg/day prednisone therapeutic dosage is permitted; prophylactic medication is allowed.
12. Any active infection requiring systemic anti-infective therapy within 14 days prior to the first administration of the Investigational Product;
13. Within 28 days prior to the first administration of the Investigational Product, the subject has undergone major surgery. In this study, major surgery is defined as a procedure requiring at least 3 weeks of postoperative recovery before being eligible to receive treatment in this study. Tumor paracentesis or lymph node incisional biopsy is permitted for enrollment.
14. Strong inhibitors or strong inducers of CYP2D6 or CYP3A were used within 2 weeks prior to the first administration of the drug.
15. Received live viral vaccine treatment within 28 days prior to the first administration of the Investigational Product; however, inactivated viral vaccines for seasonal flu and novel coronavirus are permitted;
16. Participating in another clinical trial or planning to start this study with less than 14 days since the end-of-therapy of the previous clinical trial; less than 5 half-lives since the last course of anti-tumor therapy;
17. Known to have a severe allergy to any monoclonal antibody;
18. Subjects who are not suitable for participating in this clinical study due to any clinical or laboratory abnormalities or other reasons as assessed by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2025-02-25 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
DLT | 21 days after the first dose
  The proportion of subjects experiencing dose-limiting toxicity (DLT) events in each dosage group during the DLT observation period
MTD | through study completion, an average of 12 months
  The maximum tolerated dose of HLX43 incombination with serplulimab
ORR | up to 24 weeks
  Objective response rate (ORR) (assessed by the IRRC according to the RECIST v1.1 criteria)

SECONDARY OUTCOMES:
Incidence and severity of adverse events (AEs) | from the date of the first dose to to 90 days after the last dose or the initiation of another anticancer treatment (whichever occurs first).
  severity determined according to National Cancer Institute Common Terminology Criteria for Adverse Events [NCI CTCAE] Version [v] 5.0
RP2/3D | through study completion, an average of 12 months
  RP2/3D of HLX43 combined with serplulimab in NSCLC patients
PFS | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 15 months
  Defined as the time (in months) from randomization to the first confirmed and documented progressive disease or death (whichever occurs first) as assessed by the IRRC according to the RECIST v1.1 criteria.
PFS | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 15 months
  Defined as the time (in months) from randomization to the first confirmed and documented progressive disease or death (whichever occurs first) as assessed by INV according to the RECIST v1.1 criteria.
ORR | up to 24 week
  Objective response rate (ORR) (assessed by INV according to the RECIST v1.1 criteria)
OS | From randomization to death from any cause (up to approximately 25 months)
  Overall Survival

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Hunan Provincial Cancer Hospital, Hunan, Changsha
  - Shandong Cancer Hospital, Jinan, Shangdong
  - Second Affiliated Hospital of Army Medical University, PLA, Chongqing